CLINICAL TRIAL: NCT01606696
Title: Practical Use of Higher Intensity Interval Exercise in Cardiac Rehabilitation to Improve Aerobic Fitness
Brief Title: Higher Intensity Interval Training in Cardiac Rehabilitation
Acronym: HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Steven J. Keteyian, Program Director, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HFHS-PC-HIIT
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: CAD
Keywords: CAD; cardiac rehabilitation; fitness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIIT (Experimental): Higher intensity interval training.
  Interventions: Behavioral: HIIT
- Standard intensity non-interval training (Active Comparator): Standard intensity non-interval training
  Interventions: Behavioral: Standard intensity non-interval training

INTERVENTIONS:
Behavioral: HIIT — Higher intensity interval training.
  Arms: HIIT
Behavioral: Standard intensity non-interval training — Standard intensity non-interval training.
  Arms: Standard intensity non-interval training

SUMMARY:
The purpose of this study is to compare the effect higher intensity interval exercise (HIIT) with standard intensity non-interval exercise on fitness in cardiac rehabilitation patients with CAD. Also to assess practical implementation of HIIT in cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Male or female
* Angiographic documentation of CAD

Exclusion Criteria:

* Unstable angina pectoris
* MI / PCI < 3 weeks
* CABG < 4weeks
* Exercise induced ischemia > 1mm ST depression
* LVEF < 40%
* complex ventricular arrhythmias or atrial fibrillation
* orthopedic limitations to treadmill exercise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular fitness | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Keteyian, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States